CLINICAL TRIAL: NCT05038423
Title: The 5R Shared Leadership Program in Older Adult Walking Groups: A Clustered Randomised Controlled Trial
Brief Title: The 5R Shared Leadership Program in Older Adult Walking Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Katrien Fransen, Associate professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G- 2019 02 1530
Record Dates: First submitted 2021-08-27; First posted 2021-09-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Leadership; Identification; Empowerment
Keywords: 5RS; group identification; social identification; peer leadership; identity leadership; elderly; physical activity; well-being; cohesion; walking group
MeSH Terms: conditions — Empowerment; Social Identification; Motor Activity

STUDY DESIGN:
Intervention Model Description: Clustered randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A structured 12-week group walking program (Active Comparator): Participants engaged in an evidence-based 12-week walking program.
  Interventions: Behavioral: 12-week structured walking program
- A structured 12-week group walking program + 5RS (Experimental): In addition to the 12-week group walking program, participants engaged in the 5R Shared Leadership Program, which implements a structure of shared leadership and strengthens the identity leadership skills of the appointed peer leaders.
  Interventions: Behavioral: 5R Shared Leadership Program; Behavioral: 12-week structured walking program

INTERVENTIONS:
Behavioral: 5R Shared Leadership Program — The manualised 5RS program aims to develop the leadership qualities of peer leaders by teaching them how to create, embody, advance, and embed a collective sense of 'us' in their teams. More specifically, 5RS consists of two key components that involve (1) implementing a structure of shared leadership, and (2) strengthening the identity leadership skills of the appointed peer leaders (Fransen et al., 2020).
  Fransen, K., Haslam, S. A., Steffens, N. K., Mallett, C. J., Peters, K., Mertens, N., & Boen, F. (2020). All for us and us for all: Introducing the 5R Shared Leadership Program. Psychology of Sport and Exercise, 51, 101762. https://doi.org/10.1016/j.psychsport.2020.101762 Haslam, S. A., Steffens, N. K., Peters, K., Boyce, R. A., Mallett, C. J., & Fransen, K. (2017). A social identity approach to leadership development: The 5R program. Journal of Personnel Psychology, 16(3), 113-124. https://doi.org/10.1027/1866-5888/a000176
  Arms: A structured 12-week group walking program + 5RS
Behavioral: 12-week structured walking program — Participants engaged in an evidence-based 12-week structured walking program, which aimed to enhance participants' physical activity and aerobic fitness levels based on personalised walking schedules and weekly group walks organised by the community-based meeting points.

SUMMARY:
To test the efficacy of the 5R Shared Leadership program in older adults on participants' identification with their walking group, group cohesion, walking activity, and well-being, compared to a regular group walking program, the investigators conducted a cluster randomised trial.

DETAILED DESCRIPTION:
All walking groups participated in a 12-week structured group walking program. Half of these walking groups were randomly assigned to the intervention condition and received additionally the 5R Shared Leadership Program

ELIGIBILITY:
Inclusion Criteria:

* Being part of a community-based OKRA SPORT+ meeting point that engages in the 12-week walking program

Exclusion Criteria:

* n/a

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Identity leadership | 12 weeks
  4-item Identity Leadership Inventory-Short Form
Group identification scale | 12 weeks
  To assess participants' identification with their walking group, the investigators use the 4-item group identification measure (e.g., "I am glad to be a member of this walking group."), as suggested by Doosje et al. (1995). The cognitive, evaluative, and affective aspects of identification are evaluated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree).
  Doosje B, Ellemers N, Spears R. Perceived intragroup variability as a function of group status and identification. J Exp Soc Psychol. 1995;31(5):410-36.

SECONDARY OUTCOMES:
Group cohesion | 12 weeks
  Group Environment Questionnaire - A higher score corresponds with a higher group cohesion
Well-being | 12 weeks
  Warwick-Edinburgh Mental Well-Being Scale. It comprises 14 positively phrased items (e.g., "I've been feeling good about myself") rated on a 5-point Likert scale ranging from 1 (none of the time) to 5 (all of the time). A higher score corresponds with a higher well-being
Walking activity | 12 weeks
  International Physical Activity Questionnaire - Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Fransen, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data will be shared upon publication.
Supporting Information: ICF
Time Frame: Upon publication
Access Criteria: The data will be shared together with the article following the journal recommendations.

REFERENCES:
- [Background] Fransen, K., Haslam, S. A., Steffens, N. K., Mallett, C. J., Peters, K., Mertens, N., & Boen, F. (2020). All for us and us for all: Introducing the 5R Shared Leadership Program. Psychology of Sport and Exercise, 51, 101762. https://doi.org/10.1016/j.psychsport.2020.101762
- [Derived] Fransen K, Cruwys T, Haslam C, Iserbyt P, Seghers J, Vanderlinden J, van Uffelen J, Verbaanderd E, Boen F. Leading the way together: a cluster randomised controlled trial of the 5R Shared Leadership Program in older adult walking groups. Int J Behav Nutr Phys Act. 2022 Jun 3;19(1):63. doi: 10.1186/s12966-022-01297-x. PMID 35658869